CLINICAL TRIAL: NCT06648291
Title: Telehealth Program Effectiveness in Reducing Cardiac Symptom Distress, Improving Self-care, and Enhancing Quality of Life Among Coronary Artery Disease Patients After Bypass Surgery
Brief Title: The Effectiveness of a Telehealth Program on Cardiac Symptom Distress, Self-care and Quality of Life of Patients With Coronary Artery Disease After Coronary Artery Bypass Surgery: A Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202307014RINA
Record Dates: First submitted 2024-10-06; First posted 2024-10-18 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: Telehealth; Coronary Artery Bypass Surgery
Keywords: symptoms distress; self-care; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth (Experimental): Through remote monitoring of various physiological data uploaded by the patient, immediate contact will be made when abnormal values are detected to provide individualized health education. This approach encourages the maintenance of a healthy lifestyle and facilitates early problem detection to prevent the worsening of symptoms.
  Interventions: Device: QOCA EKG Device
- Usual care (Placebo Comparator): Provide post-operative education on the day of discharge and follow up with a phone call one week after discharge to check on the patient.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: QOCA EKG Device — The investigators scheduled telephone interviews every three days to encourage and monitor the development of good self-health care behaviors by: (1) asking about daily blood pressure, weight, and lower extremity edema; (2) providing medication counseling, as well as exercise and dietary hygiene recommendations; (3) offering wound care guidance; (4) advising on the proper use of wounds; (5) advising on avoiding cardiac risk factors such as smoking and secondhand smoke; and (6) following up on physical status at outpatient clinics and assisting with referrals to relevant clinics, such as nutrition or rehabilitation, based on the patient's condition. A QOCA portable electrocardiogram (ECG) measurement device will be provided for patients to use at home. In the event of abnormal physiological values, the investigator will contact the patient to assess his or her medical status and provide 24-hour online counseling.
  Arms: Telehealth
Other: Usual Care — Provide post-operative education on the day of discharge and follow up with a phone call one week after discharge to check on the patient.
  Arms: Usual care

SUMMARY:
The goal of this randomized trial is to compare the outcomes of a telehealth program with conventional discharge care for patients aged 18 years and older with coronary artery disease following coronary artery bypass surgery. The main question it seeks to answer are:

1. To investigate whether there is a difference in symptom distress between patients with coronary artery disease receiving a telehealth program after CABG (experimental group) and those receiving usual care (control group).
2. To examine whether there is a difference in self-care behaviors between patients with coronary artery disease receiving a telehealth program after CABG (experimental group) and those receiving usual care (control group).
3. To investigate whether there is a difference in the quality of life of patients with coronary artery disease receiving a telehealth program (experimental group) after CABG compared to those receiving usual care (control group).

Participants will be randomly assigned to one of two groups: either a telehealth program or usual care. The Symptom Distress, Self-Care, and SF-12 Quality of Life Questionnaire will be used to assess and track symptom distress, self-care, and quality of life two days prior to discharge, during the first post-discharge visit (days 7 to 10), and in the fourth week post-discharge. The aim is to alleviate symptom distress in patients returning home after coronary artery bypass surgery, enhance self-care behaviors, and ultimately improve quality of life. This study seeks to maximize the benefits of a telehealth program, establishing it as an important care strategy for future integration with hospital-based care.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of a telehealth program for patients discharged after coronary artery bypass surgery, specifically examining whether it reduces symptom distress, improves self-care skills, and enhances quality of life compared to usual care.

Background:

Cardiovascular diseases (CVD) contribute substantially to global mortality rates and have consistently ranked as the second leading cause of death in Taiwan for many years.Coronary artery bypass graft (CABG) is an important and common surgical procedure for treating cardiovascular disease. However, one in four patients who undergo CABG suffers from postoperative complications, including pain, wound infections, and sleep disturbances, which can further impact their quality of life. Some of these symptoms may last from weeks to months, and if left unresolved, they may hinder the patient's recovery and increase the risk of death. Additionally, shorter hospital stays make it more challenging for patients to transition from hospital to home and adjust to changes in their lives, which can lead to poorer self-care behaviors and worsen complications such as heart failure, wound infections, and cardiac arrhythmia, seriously affecting their quality of life.

Telehealth refers to the use of communication technology, electronic medical equipment, and professional medical technology to provide the public with a wider range of medical care services in familiar community or home environments, facilitating local aging. Its functions and benefits encompass four major dimensions:

1. . Physiological information monitoring: This includes the transmission, storage, and utilization of data such as blood pressure, blood glucose, and pulse. The consolidated data can serve as a basis for adjusting medication.
2. . Contact and coordination of care services: This involves emergency responses from the patient side, monitoring of abnormal signals, and reminders for follow-up visits.
3. . Assistance in self-health management: This entails monitoring changes in the patient's daily physiological parameters and encouraging self-management and tracking, including exercise, medication, diet, and maintaining a healthy lifestyle.
4. Video consultations: Nurses and patients can communicate over long distances to achieve effective monitoring and control, breaking geographical constraints. This allows for customized health consultations and guidance, as well as emotional support.

International literature confirms that telehelth services can reduce healthcare costs, emergency room visits, readmission rates, and mortality rates.

Study Design and Interventions:

The study adopts an open-label, two-arm, parallel-group randomized controlled design. Participants will be randomly assigned into one of two groups:

Experimental group: Telehealth program Control group:Usual care (Routine hospital discharge care) Experimental Group: Patients will be discharged from the hospital to telehealth program with the following interventions.

Telephone interviews were arranged every three days by the investigator, who had more than 10 years of experience in case management practice and was certified as a cardiovascular and diabetes health teacher. The main purpose of the telephone interviews was to encourage and supervise the patients to develop good self-health care behaviors, which included: (1) asking about the daily blood pressure, weight, and edema of the lower limbs (2) providing medication counseling, and exercise and dietary hygiene (3) wound care advice (4) providing advice on the use of wounds, and (5) providing advice on the use of wounds, and (6) providing advice on the use of wounds, and (7) providing advice on the use of wounds. Wound care guidance (4) Avoidance of heart disease risk factors such as smoking and second-hand smoke (5) Tracking of physical condition at the time of outpatient visit and assisting in referral to relevant outpatient clinics such as nutrition or rehabilitation clinics according to the patient's condition. In addition to this, a set of QOCA portable electrocardiogram (ECG) measuring device will be provided for use at home. During the hospitalization period, we will ask the vendor to assist in installing the ECG software on the patient's cell phone, instructing the patient on how to operate the device and repeat the instructions until the patient is able to operate it by themselves. Repeat the instructions until the patient is able to operate the device on his/her own, and bring back a manual with instructions for operation, informing the patient that the frequency of measurements should be once in the morning and once in the evening, but if he/she has chest congestion, he/she can upload the measurements at any time, and send the website address of the center's platform and the operation procedures to the patient by SMS, asking him/her to enter the daily physiological values of blood pressure and blood glucose, and the researcher will contact him/her to assess his/her medical condition when there are abnormalities in the cardiac rhythms, blood pressure, or blood glucose, and provide 24-hour online counseling services. Provide 24-hour online counseling service to detect problems as early as possible and handle them immediately to avoid deterioration of their symptoms.

In the control group, subjects were given routine discharge counseling and telephone follow-up within 7 days of discharge.

Study Duration and Data Collection: The study will last 4 weeks for each participant. Data will be collected from hospital records, patient self-reports and questionnaire scales. Measured outcomes will include:

Primary outcome: degree of improvement in symptom distress, self-care ability, and quality of life.

Secondary Outcome: Physiologic data (e.g., blood pressure, heart rate, and weight).

Randomization and Recruitment: Participants will be recruited from cardiology wards according to the inclusion criteria (patients undergoing first time coronary artery bypass surgery). Randomization will be randomly coded, with numbers placed in envelopes numbered from 1 to 160, which will be self-administered, with odd-numbered subjects assigned to the experimental group and even-numbered subjects assigned to the control group.

Significance: This study will evaluate the effectiveness of a telehealth program compared with usual care, with the goal of improving telehealth service quality. The intervention is expected to reduce symptom distress, strengthen self-care behaviors, and improve quality of life among patients recovering at home after coronary artery bypass surgery. Ultimately, the findings may support telehealth as an essential care strategy for integration into future hospital-based services.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≧18 years old
* Ability to read and answer questionnaires in Chinese.
* After coronary artery bypass surgery (CABG)
* Able to install and download the QOCA ECG software on their cell phones

Exclusion Criteria:

* Inability to communicate effectively and cognitive impairment
* Unable to take care of themselves or are physically disabled.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2025-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chih-Hui Shih, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) due to concerns about maintaining participant privacy and confidentiality. The study involves sensitive health information, and ensuring the protection of participant identity is a priority.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telehealth | Usual Care
Started | 80 | 80
Completed | 78 | 76
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — difficulty using the equipment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telehealth | Usual Care | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is reported as mean and standard deviation (years)
  years | 67.06 (9.06) | 65.3 (10.10) | 66.19 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex is reported as the number of participants in each category (female and male).
  Participants
    Female | 15 | 8 | 23
    Male | 65 | 72 | 137
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Symptom Distress Score
Description: Cardiac symptom distress was assessed using the Cardiac Symptom Survey (CSS). The CSS consists of 10 items assessing common cardiac-related symptoms, including angina, shortness of breath, fatigue, depression, sleep disturbance, incisional pain, leg edema, palpitations, anxiety, and loss of appetite.
  For each symptom, participants rated symptom frequency and severity on separate 0-10 scales (0 = none, 10 = extremely severe). A mean score for each symptom was calculated by averaging the frequency and severity ratings. The total cardiac symptom distress score was obtained by summing the mean scores of all 10 symptoms, with higher scores indicating greater symptom distress.
Time Frame: Assessed at three time points: baseline (2 days before hospital discharge), 7-10 days after hospital discharge, and 4 weeks after hospital discharge
Population: A total of 160 participants were randomized. Six participants did not complete follow-up assessments due to equipment issues, need for ECG monitoring, loss to follow-up, or death. Therefore, outcome analyses were conducted on 154 participants (78 in the intervention group and 76 in the control group
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Usual Care: Participants in the usual care group received standard postoperative care according to routine hospital practice. This included postoperative education provided on the day of discharge and a routine follow-up phone call approximately one week after discharge to assess the patient's condition. No telehealth monitoring or additional remote support was provided.
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 78 | 76
scores on a scale
  Baseline (2 days before hospital discharge) | 15.24 (10.61) | 12.84 (8.94)
  7-10 days after hospital discharge | 12.81 (11.57) | 11.87 (10.68)
  4 weeks after hospital discharge | 8.1 (8.07) | 11.76 (12.21)

2. Secondary Outcome: Self-care Behavior Score
Description: Self-care behavior was assessed using the Self-Care Behavior Scale developed for patients undergoing coronary artery bypass graft surgery. The scale consists of 16 items assessing engagement in self-care activities and control of cardiovascular risk factors. Each item is rated on a 4-point Likert scale (1 = never to 4 = always). Item scores are summed to yield a total score ranging from 16 to 64, with higher scores indicating better self-care behavior. Units of measure: scores on a scale.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | Telehealth
Number analyzed (Participants) | 76 | 78
scores on a scale
  Baseline (2 days before hospital discharge) | 50.57 (8.59) | 49.60 (8.4)
  7-10 days after hospital discharge | 58.59 (3.93) | 57.16 (5.53)
  4 weeks after hospital discharge | 59.94 (4.16) | 56.93 (6.31)

3. Secondary Outcome: SF-12 Physical Component Summary (PCS)
Description: Health-related quality of life was assessed using the 12-Item Short Form Health Survey (SF-12, Version 1). The Physical Component Summary (PCS) score reflects physical aspects of health-related quality of life and is derived from the physical health-related domains of the SF-12. PCS scores are standardized on a 0-100 scale, with higher scores indicating better physical health status. Units of measure: scores on a scale.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 78 | 76
scores on a scale
  Baseline (2 days before hospital discharge) | 30.48 (5.75) | 32.49 (6.96)
  7-10 days after hospital discharge | 35.38 (8.94) | 35.21 (8.35)
  4 weeks after hospital discharge | 37.92 (8.53) | 37.36 (8.88)

4. Secondary Outcome: SF-12 Mental Component Summary (MCS)
Description: Health-related quality of life was assessed using the 12-Item Short Form Health Survey (SF-12, Version 1). The Mental Component Summary (MCS) score reflects the mental and emotional aspects of health-related quality of life, including vitality, social functioning, role limitations due to emotional problems, and mental health. The MCS score is a norm-based summary score derived from weighted combinations of SF-12 item responses according to standard scoring algorithms. Scores are standardized on a 0-100 scale, with higher scores indicating better mental health status. Units of measure: scores on a scale.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Telehealth | Usual Care
Number analyzed (Participants) | 78 | 76
scores on a scale
  Baseline (2 days before hospital discharge) | 47.96 (10.71) | 49.27 (10.47)
  7-10 days after hospital discharge | 48.28 (9.63) | 50.36 (10.04)
  4 weeks after hospital discharge | 50.53 (9.29) | 50.18 (10.28)

ADVERSE EVENTS:
Time Frame: From baseline (hospital discharge) up to 4 weeks after hospital discharge.
Description: Adverse events were assessed through routine follow-up and review of medical records. Serious adverse events, including all-cause mortality, were recorded for all enrolled participants in accordance with ClinicalTrials.gov definitions. The relationship between adverse events and the study intervention was determined by the study investigators.
Arm/Group | Telehealth | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/78 | 1/76
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/76
Other Adverse Events (participants affected / at risk) | 0/78 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT06648291/Prot_SAP_000.pdf